CLINICAL TRIAL: NCT00423683
Title: A Randomized Control Trial of Anticoagulation and Inferior Vena Cava Filters in Cancer Patients With A Venous Thromboembolism
Brief Title: Anticoagulation and Inferior Vena Cava Filters in Cancer Patients With a Venous Thromboembolism
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study accrual stopped due to poor accrual.
Sponsor: Northwell Health (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Daniel Budman, Interim Chief, Division of Oncology, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB # 06-034
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Results first posted 2016-05-03 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-05

CONDITIONS: Cancer; Thromboembolism
Keywords: Cancer; thromboembolism
MeSH Terms: conditions — Neoplasms; Thromboembolism | interventions — Fondaparinux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1- Arixtra Alone (Experimental): Arixtra Alone
  Interventions: Drug: Arixtra alone
- 2 Arixtra+ filter (Active Comparator): Arixtra + filter
  Interventions: Device: Arixtra + filter

INTERVENTIONS:
Drug: Arixtra alone — Arixtra subq injection 5mg dose (dose also dependent upon size and age of pt)
  Other Names: Arixtra
  Arms: 1- Arixtra Alone
Device: Arixtra + filter — Arixtra as daily injections similar to arm I and placement of Inferior Vena Cava (IVC) filter.
  Other Names: IVC filter and Arixtra
  Arms: 2 Arixtra+ filter

SUMMARY:
The development of clots is a potentially deadly complication in many cancer patients. The current optimal treatment is unknown. Evidence supporting the effectiveness of the use of Inferior Vena Caval Filters is lacking. This study will compare the two standard of care treatment options: anticoagulation with or without a inferior vena cava filter. The anticoagulation medication chosen will be Arixtra and it will be given once a day as an injection. Patients will be called at various intervals to monitor their signs and symptoms of new thromboembolisms.

DETAILED DESCRIPTION:
The development of clots is a potentially deadly complication in many cancer patients. The current optimal treatment is unknown. Evidence supporting the effectiveness of the use of Inferior Vena Caval Filters is lacking. This study will compare the two standard of care treatment options: anticoagulation with or without an inferior vena cava filter. The anticoagulation medication chosen will be Arixtra and it will be given once a day as an injection. Patients will be called at various intervals to monitor their signs and symptoms of new thromboembolisms. Patients will be equally randomized to receive either Arixtra with or without placement of an Inferior Vena Cava (IVC) filter. Fifty three patients are expected to be enrolled in each arm. Patients will be monitored for 90 days after study enrollment. Monitoring will include telephone calls and physician visits and repeat radiologists if the patient is symptomatic of a Deep Vein thrombosis (DVT). This will also include completion of a quality of life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of cancer.
* The disease may be a solid tumor, Lymphoma or Multiple Myeloma. Pathology reports will be documented in the patient's chart and included in the data.
* Age > 18 years
* An acute, radiographically confirmed, de novo Deep Vein Thrombosis (DVT) or Pulmonary Embolism (PE)
* No past medical history of a prior thrombus or known thrombophilia

Exclusion Criteria

* Patients are not eligible for this study if they receive therapeutic doses of any heparin for more than 72 hours before randomization 31.
* Already receiving oral anticoagulant therapy 31.
* Severe renal impairment, calculated using the Cockcroft-Gault formula, defined as a creatinine clearance <30 mL/min 31.
* Platelet count of less than 50,000 per cubic millimeter
* Bleeding from the gastrointestinal tract that requires blood transfusion (s), intracranial bleeding or retroperitoneal bleeding.
* An indication for thrombolysis
* Allergy to iodine
* Hereditary thrombophilia
* Pregnancy
* Likelihood of noncompliance
* It is contraindicated to anticoagulate patients with brain metastasis secondary to melanoma, choriocarcinoma, renal cell and medullary thyroid carcinoma. If these patients have a Venous Thromboembolism (VTE), it is standard of care for these patients to have a CT of their head to evaluate if there is metastasis to the brain before they are anticoagulated 38. If these patients do have brain metastasis, they will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myra Barginear, MD, Principal Investigator — North Shore University Hospital Monter Cancer Center; Daniel R. Budman, MD, Principal Investigator — North Shore University Hospital Monter Cancer Center
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment was slowed due to newly approved medications so study was stopped early.
Groups:
- 2 Arixtra+ Filter: Arixtra subq injection + IVC filter
- 1-Arixtra Alone: Arixtra treatment without inferior vena cava filter
Period: Overall Study
Arm/Group | 2 Arixtra+ Filter | 1-Arixtra Alone
Started | 31 | 33
Completed | 30 | 33
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1- Arixtra Alone: Arixtra treatment without inferior vena cava filter
- Total: Total of all reporting groups
Arm/Group | 2 Arixtra+ Filter | 1- Arixtra Alone | Total
Number analyzed (Participants) | 31 | 33 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 12 | 33
  >=65 years | 10 | 21 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (2) | 67 (14) | 65 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 24 | 40
  Male | 15 | 9 | 24
Region of Enrollment [Number; unit: participants]
  United States | 31 | 33 | 64

OUTCOME MEASURES:

1. Primary Outcome: Adverse Outcomes
Description: Rates of VCF complications, bleeding, and recurrent or residual DVTs or PEs
Time Frame: 3 years or until death
Measure: Number; unit: percentage of participants
Arm/Group | Arixtra | Arixtra and Filter
Number analyzed (Participants) | 33 | 31
percentage of participants | 15.2 | 16.1

2. Secondary Outcome: Overall Survival
Time Frame: 3 years or until death
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm 1 Arixtra | Arm 2 Arixtra + IVC Filter
Number analyzed (Participants) | 33 | 31
days | 493 [141 to 744] | 266 [118 to 426]

3. Secondary Outcome: Resolution of DVT
Time Frame: 3 years or until death
Population: 33 participants contributed 59 DVT sites in Arm 1; 31 participants contributed 48 DVT sites in Arm 2. Unit of analysis was DVT sites
Measure: Number; unit: percentage of DVT sites
Units Other Than Participants: DVT sites
Arm/Group | Arm 1 Arixtra | Arm 2 Arixtra + IVC Filter
Number analyzed (Participants) | 33 | 31
Number analyzed (DVT sites) | 59 | 48
percentage of DVT sites | 61.0 | 37.5

4. Secondary Outcome: Resolution of PE
Time Frame: 3 years or until death
Population: 33 participants contributed 25 PE sites in Arm 1; 31 participants contributed 18 PE sites in Arm 2. Unit of analysis was PE sites
Measure: Number; unit: percentage of PE sites
Units Other Than Participants: PE sites
Arm/Group | Arm 1 Arixtra | Arm 2 Arixtra + IVC Filter
Number analyzed (Participants) | 33 | 31
Number analyzed (PE sites) | 25 | 18
percentage of PE sites | 32.0 | 66.7

ADVERSE EVENTS:
Groups:
- Arixtra Alone: Arixtra anti coagulation alone
Arm/Group | 2 Arixtra+ Filter | Arixtra Alone
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/33
Other Adverse Events (participants affected / at risk) | 0/31 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less